CLINICAL TRIAL: NCT05562323
Title: Characterization of Vaccine-induced Responses Against Monkeypox (MoVIHvax) An Observational Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other); BCN Checkpoint (Industry)
Responsible Party: Sponsor
Other Study IDs: MoVIHvax
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Monkeypox
Keywords: Monkeypox vaccine; Immune responses; HIV
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples: PBMC, plasma and whole blood in PaxGene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MKP vaccination for pre-exposure prophylaxis (HIV positive): HIV positive individuals who receive MKP vaccination for pre-exposure prophylaxis
- MKP vaccination for pre-exposure prophylaxis (seronegative individuals): HIV seronegative individuals who receive MKP vaccination for pre-exposure prophylaxis

SUMMARY:
This observational study has been designed to characterize humoral and cellular immune responses after vaccination against monkeypox (MKP) in HIV positive and negative individuals at high risk of MKP infection during the vaccination campaign in the current monkeypox outbreak.

DETAILED DESCRIPTION:
Of the 23,837 cases of monkeypox reported in the European Region of the WHO, 7.037 have been identified in Spain, according to the National Epidemiological Surveillance Network (RENAVE). Most of diagnosed individuals are men born in Spain, being nearly 40% HIV positive. The clinical evolution was satisfactory, although 3-7% of cases required hospitalization.

Given the limited number of available doses of the MVA-BN vaccine, it has been recently approved its use as a single intradermal dose. However, this posology can be more reactogenic than subcutaneous injection and there is limited data on its immunogenicity and effectiveness in people living with HIV (PLWH), which account for about half of the monkeypox cases in the current outbreak.

The present observational study has been designed to investigate the humoral and cellular immune responses following monkeypox vaccination in PLWH.

ELIGIBILITY:
Inclusion Criteria:

1. Adult individuals of ≥18 years old.
2. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the trial.
3. Has understood the information provided and capable of giving informed consent.

Exclusion Criteria:

1. Participant has any medical condition and/or finding that in the investigator opinion might increase participant risks, interfere with the study or impair interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 individuals who have been/will be vaccinated against MKP as pre-exposuire profilaxis following the National Vaccination Plan (40-50/50-60% of HIV negative and HIV positive individuals)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with detectable anti-orthopox antibodies | Between day 29 - 90
  Proportion of participants with detectable anti-orthopox antibodies at 29 - 90 days following first MVA-BN vaccination
Quantification of anti-orthopox antibodies | Between day 29 - 90
  Quantification of anti-orthopox antibodies at 29 - 90 days following first MVA-BN vaccination

SECONDARY OUTCOMES:
Changes of the immunogenicity after the first vaccine dose | Between day 29 - 90 and between 150-180 (after the first dose) and between 29 - 90 and between 150-180 (after the second dose if applicable)
  The geometric mean fold rise (GMFR) in anti-orthopox antibody titers from baseline to Day 29-90 and 150-180 after the first dose of MVA-BN and to 29-90 and 150-180 after the second dose (if applicable)
To compare immunogenicity between HIV negative and HIV positive individuals | Between day 29 - 90 and between 150-180 (after the first dose) and between 29 - 90 and between 150-180 (after the second dose if applicable)
  To compare the GMFR between HIV negative and HIV positive individuals
Neutralization capacity of anti-orthopox antibodies | Between day 29 - 90 and between 150-180 (after the first dose) and between 29 - 90 and between 150-180 (after the second dose if applicable)
  Neutralization titers measured as the reciprocal dilution inhibiting 50% of the infection (ID50) will be reported using a live virus assay (VNA) to measure cytopathic effect in Vero E6 cells after the first dose of MVA-BN.
To compare neutralization capacity between HIV negative and HIV positive individuals | Between day 29 - 90 and between 150-180 (after the first dose) and between 29 - 90 and between 150-180 (after the second dose if applicable)
  To compare ID50 between HIV negative and HIV positive individuals

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - BCN Checkpoint, Barcelona, Barcelona
  - VALLE HEBRÓN HOSPITAL/Centro Salud Internacional y Enfermedades Transmisibles Drassanes, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No